### The GlaxoSmithKline group of companies

| Division | : | Worldwide Development |
|------------------|---|-----------------------------------|
| Information Type | : | Reporting and Analysis Plan (RAP) |

| Title | : | A 2-Part, Phase I, Single-Dose, 3-Period Crossover Relative<br>Bioavailability Study of a Pediatric TRIUMEQ Dispersible<br>Tablet and Pediatric Dolutegravir and Lamivudine<br>(DTG/3TC) Fixed Dose Combination Dispersible Tablet<br>Formulations as Compared With Adult Tablets in Healthy<br>Volunteers |
|---|---|---|
| Compound Number | : | GSK1349572+GR109714+GI265235 (GSK2619619) and GSK1349572+GR109714 (GSK3515864) |
| Effective Date | : | 25-APR-2018 |

### **Description:**

- The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Study Report for Protocol 205894.
- This RAP is intended to describe the safety, tolerability, and pharmacokinetic (PK) analyses required for the study.
- This RAP will be provided to the study team members to convey the content of the Statistical Analysis Complete (SAC) deliverable.

#### **Author's Name and Functional Area:**

| PPD | 25-APR-2018 |
|---|---|
| Biostatistician II (Biostatistics, Early Development Services, PPD) | 23-APK-2018 |
| PPD | 25 ADD 2019 |
| Pharmacokineticist (Biostatistics, PPD) 25-APR-2018 | |

### Approved by:

| PPD | | |
|--------------------|---------------------------------|-------------|
| Principal Statisti | cian (Clinical Statistics, GSK) | 25-APR-2018 |

Copyright 2018 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

# The GlaxoSmithKline group of companies

# Approved by:

| Approver | Date | Approval Method |
|-------------------------------------|--------------|-----------------|
| PPD | 18-APR-2018 | e-mail |
| Global Clinical Development Manager | 16-A1 K-2016 | |
| PPD | 10 ADD 2010 | e-mail |
| Director, Clinical Development | 19-APR-2018 | |
| PPD | 19-APR-2018 | e-mail |
| Director, Clinical Pharmacology | 19-APK-2018 | |
| PPD | 10 ADD 2010 | e-mail |
| SERM Manager | 19-APR-2018 | |
| PPD | 10 ADD 2010 | e-mail |
| Principal Programmer/Analyst | 19-APR-2018 | |
| PPD | 10 ADD 2010 | e-mail |
| Principal Data Manager | 19-APR-2018 | |

# **TABLE OF CONTENTS**

| | | | | | PAGE |
|---|---|---|---|---|---|
| 1. | REPO | RTING & | ANALYSIS | PLAN SYNPOSIS | 5 |
| 2. | STIMM | IADV OE I | ZEV DD∩T | OCOL INFORMATION | 0 |
| ۷. | 2.1. | | | tocol Defined Statistical Analysis Plan | |
| | 2.1. | | | and Endpoint(s) | |
| | 2.3. | | | and Endpoint(s) | |
| | 2.4. | | | es | |
| 3. | PLANI | NED ANA | LYSES | | 12 |
| | 3.1. | Final Ana | alyses | | 12 |
| 4. | ΔΝΔΙΝ | VSIS POP | ΙΙΙ ΔΤΙΩΝΟ | S | 13 |
| т. | 4.1. | | | | |
| _ | | | | | 10 |
| 5. | | | | DATA ANALYSES AND DATA HANDLING | 14 |
| 6. | | | | ALYSES | |
| | 6.1. | Overview | of Planne | d Analyses | 15 |
| 7. | PRIMA | ARY STAT | ISTICAL A | NALYSES | 16 |
| | 7.1. | Pharmac | okinetic Ar | nalyses | 16 |
| | | 7.1.1. | | of Planned Pharmacokinetic Analyses | |
| | | 7.1.2. | | centration Measures | |
| | | 7.1.3. | | kinetic Parameters | |
| | | | 7.1.3.1. | 5 | 16 |
| | | | 7.1.3.2. | Statistical Analysis of Pharmacokinetic | |
| | | | | Parameters | |
| | | 7.1.4. | | nalysis | |
| | | | 7.1.4.1. | Overview of Planned Analyses | 19 |
| 8. | SECO | NDARY S | TATISTICA | AL ANALYSES | 20 |
| | 8.1. | Safety A | nalyses | | 20 |
| | 8.2. | • | • | es | |
| 9. | REFE | RENCES. | | | 22 |
| 10 | A DDEI | NDICES | | | 22 |
| 10. | 10.1. | | | Events | |
| | 10.1. | 10.1.1. | Protocol D | Defined Screening Assessments for Parts 1 and | |
| | | | | | 24 |
| | | 10.1.2. | | Defined Time and Events for Parts 1 and 2 | |
| | 10.2. | | | ent States and Phases | |
| | | 10.2.1. | | t States | |
| | | | | Treatment States for Safety Data | 27 |
| | | | 10.2.1.2. | Treatment States for Event Data (e.g. AEs, | ^ <del>-</del> |
| | 10.0 | | , 2, D-t- D | Concomitant Medications) | |
| | 10.3. | | | isplay Standards & Handling Conventions | |
| | | 10.3.1. | Study ITE | atment & Sub-group Display Descriptors | ∠ŏ |

| | 10.3.2. | Baseline D | Definition & Derivations | . 29 |
|---|---|---|---|---|
| | | 10.3.2.1. | Baseline Definitions | .29 |
| | | 10.3.2.2. | Derivations and Handling of Missing Baseline | |
| | | | Data | .29 |
| | 10.3.3. | Reporting | Process & Standards | |
| 10.4. | Appendix | | I and Transformed Data | |
| | 10.4.1. | | | |
| | 10.4.2. | Study Pop | ulation | .32 |
| | 10.4.3. | • | | |
| 10.5. | Appendix | ς 5: Premat | ure Withdrawals & Handling of Missing Data | .34 |
| | 10.5.1. | | Withdrawals | |
| | 10.5.2. | Handling of | of Missing Data | .34 |
| | | 10.5.2.1. | Handling of Missing Dates | .34 |
| | | 10.5.2.2. | Handling of Partial Dates | .35 |
| 10.6. | Appendix | 6: Values | of Potential Clinical Importance | .36 |
| | 10.6.1. | ECG | | . 36 |
| | 10.6.2. | | 3 | |
| 10.7. | Appendix | | Comparisons & Multiplicity | |
| | 10.7.1. | | of Multiple Comparisons & Multiplicity | .37 |
| 10.8. | | | Checking and Diagnostics for Statistical | |
| 10.9. | • • | | viations & Trade Marks | |
| | 10.9.1. | | ons | |
| | | | (S | |
| 10.10. | | | Data Displays | |
| | | | mple Shell Referencing | |
| | | | e [Priority] | |
| | | | ulation Tables | |
| | | | ples | |
| | | | kinetic Tables | |
| | | | kinetic Figures | |
| | | | y Tables | |
| | | | gs | |
| | | | n-ICH) Listings | |
| 10.11. | Appendix | ر 11: Examı | ole Mock Shells for Data Displays | .54 |

# 1. REPORTING & ANALYSIS PLAN SYNPOSIS

| Overview | Key Elements of the RAP |
|---|---|
| Purpose | The purpose of this reporting and analysis plan (RAP) is to describe any planned analyses and output to be included in the clinical study report for Protocol 205894. |
| Protocol | This RAP is based on the original protocol (Dated: 18/JAN/2018) of study 205894 (GlaxoSmithKline Document Number. 2017N330422_00). |
| Primary | Part 1: |
| Objective | To compare the relative bioavailability (BA) of dolutegravir (DTG), abacavir (ABC), and lamivudine (3TC) administered as pediatric TRIUMEQ dispersible tablets with the conventional adult TRIUMEQ tablet (reference) administered as direct-to-mouth when: |
| | Pediatric TRIUMEQ dispersible tablets are administered as a dispersion and taken immediately |
| | Pediatric TRIUMEQ dispersible tablets are administered as direct to-mouth. |
| | Part 2: |
| | To compare the relative BA of DTG and 3TC administered as pediatric DTG/3TC dispersible tablets with the conventional adult DTG and 3TC tablets (reference) administered as direct-to-mouth when: |
| | Pediatric DTG/3TC dispersible tablets are administered as a dispersion and taken immediately |
| | Pediatric DTG/3TC dispersible tablets are administered as direct-to-mouth |
| Primary | Parts 1 and 2: |
| Endpoint | Plasma DTG, ABC (Part 1 only), and 3TC: |
| | <ul> <li>Area under the plasma concentration-time curve (AUC) from time of dose<br/>extrapolated to infinite [AUC(0-∞)], AUC from time of dose to last measurable<br/>concentration [AUC(0-t)], and maximum observed concentration (Cmax).</li> </ul> |
| Secondary | Part 1: |
| Objectives | To compare the single-dose pharmacokinetics (PK) of DTG, ABC, and 3TC administered as pediatric TRIUMEQ dispersible tablets with the conventional adult TRIUMEQ tablets (reference) administered as direct-to-mouth when: |
| | Pediatric TRIUMEQ dispersible tablets are administered as a dispersion and taken immediately |
| | Pediatric TRIUMEQ dispersible tablets are administered as direct to-mouth |
| | To evaluate the safety and tolerability of DTG, ABC, and 3TC administered as pediatric TRIUMEQ dispersible tablets as compared with conventional adult TRIUMEQ tablet (reference) administered as direct-to-mouth |

| Overview | Key Elements of the RAP |
|---|---|
| | Part 2: |
| | <ul> <li>To compare the single-dose PK of DTG and 3TC administered as pediatric<br/>DTG/3TC dispersible tablets, with the conventional adult DTG and 3TC tablets<br/>(reference) administered as direct-to-mouth when:</li> </ul> |
| | <ul> <li>Pediatric DTG/3TC dispersible tablets are administered as a dispersion and<br/>taken immediately</li> </ul> |
| | <ul> <li>Pediatric DTG/3TC dispersible tablets are administered as direct to-mouth</li> </ul> |
| | <ul> <li>To evaluate the safety and tolerability of DTG and 3TC administered as<br/>pediatric DTG/3TC dispersible tablets as compared with the conventional adult<br/>DTG and 3TC tablets (reference) administered as direct-to-mouth</li> </ul> |
| Secondary | Parts 1 and 2: |
| Endpoints | Plasma DTG, ABC (Part 1 only) and 3TC: |
| | <ul> <li>AUC from time of dose to 24 hours [AUC(0-24)], time to maximum concentration (Tmax), time of last quantifiable concentration (Tlast), apparent oral clearance (CL/F), apparent volume of distribution (VZ/F), observed concentration at 24 hours postdose (C24), last observed quantifiable concentration (Ct), and terminal elimination phase half-life (t½),</li> </ul> |
| | Plasma DTG: lag time for absorption (tlag) |
| | <ul> <li>Safety and tolerability parameters for adverse events (AEs)/serious adverse<br/>events (SAE), observed and change from baseline clinical laboratory<br/>assessments, electrocardiogram (ECG), and vital signs</li> </ul> |
| Exploratory | Parts 1 and 2: |
| Objective | To evaluate the palatability of the dispersible tablets |
| Exploratory | Parts 1 and 2: |
| Endpoint | Palatability questionnaire |
| Study<br>Design | <ul> <li>This study will be conducted as a 2-part, open-label, single-dose, 3-period, randomized, crossover study to compare the relative BA of pediatric TRIUMEQ dispersible tablets with an adult TRIUMEQ conventional tablet formulation (Part 1) and of pediatric DTG/3TC dispersible tablets with adult DTG and 3TC conventional tablets formulation (Part 2) in healthy volunteers under fasted conditions. Prior to dosing on Day 1 of Period 1 in each part, participants will be randomized to 1 of 6 treatment sequences (ABC, BCA, CAB, ACB, BAC, or CBA in Part 1; DEF, EFD, FDE, DFE, EDF, or FED in Part 2) and will receive a single dose of each of the 3 treatments administered as 1 treatment per period. Parts 1 and 2 of the study are independent of one another and may be run in parallel.</li> <li>Treatments are defined below:</li> </ul> |

| Overview | ey Elements of the RAP | |
|---|---|---|
| | Part 1 | |
| | Treatment A: Adult TRIUMEQ (DTG 50 mg/ABC 600 mg/3TC 300 mg, 1 conventional tablet) administered as direct-to-mouth (reference) | |
| | Treatment B: Pediatric TRIUMEQ (DTG 5 mg/ABC 60 mg/3TC 30 mg, 10 dispersible tablets) administered as a dispersion and taken immediately (tes | st) |
| | Treatment C: Pediatric TRIUMEQ (DTG 5 mg/ABC 60 mg/3TC 30 mg, 10 dispersible tablets) administered as direct-to-mouth (test). | |
| | Part 2 | |
| | Treatment D: Adult DTG (50 mg, 1 conventional tablet) and adult 3TC (300 mg 1 conventional tablet) administered as direct-to-mouth (reference) | J, |
| | Treatment E: Pediatric DTG/3TC (DTG 5 mg/3TC 30 mg, 10 dispersible tablets administered as a dispersion and taken immediately (test) | 3) |
| | Treatment F: Pediatric DTG/3TC (DTG 5 mg/3TC 30 mg, 10 dispersible tablets administered as direct-to-mouth (test) | s) |
| Planned<br>Analyses | Plasma DTG, ABC (Part 1 only), and 3TC concentration-time data will be analyzed by non-compartmental methods with Phoenix WinNonlin Version 6.4 or higher. Calculations will be based on the actual sampling times recorded during the study. From the plasma concentration-time data, the following PK parameters will be determined, as data permit: Cmax, Tmax, Tlast, AUC(0-t), AUC24, AUC(0-∞), t1/2, tlag (DTG only), C24, Ct, Vz/F, and CL/F. | <b>.</b> |
| | Pharmacokinetic data for each part will be listed and may be presented in graphical form, and will be summarized descriptively. All PK data will be stored in the Archives, GlaxoSmithKline R&D. | d |
| | The primary PK parameters for DTG, ABC (Part 1 only), and 3TC in Part 1 (AUC[0-∞], AUC[0-t], and Cmax) will be loge-transformed and separately analyzed using a mixed effects model with fixed-effect terms for Period, Treatment, and Treatment Sequence for each treatment comparison. Participant will be nested within Treatment Sequence and treated as a random effect in the model. Point estimates and their associated 90% CIs will be constructed for the differences in PK parameter values between test and reference treatments. The point estimates and their associated 90% CIs will then be back transformed to provide point estimates and 90% CIs for the ratio of PK parameters from test and reference treatments. | |
| | Safety data for each part will be presented in tabular format and summarized descriptively according to GSK's Integrated Data Standards Library (IDSL) standards. No formal statistical analysis of the safety data will be conducted. | |
| | Palatability questionnaire variables for each part will be summarized descriptively. | |
| Analysis<br>Populations | All Participants Population: all participants who receive at least 1 dose of study medication. This population will be used for all demographic and safety | у |

| Overview | Key Elements of the RAP |
|---|---|
| | summaries |
| | PK Population: participants in the 'All Participants' population for whom a PK sample was obtained and who had evaluable PK assay results. PK samples that may be affected by protocol deviations will be reviewed by the study team to determine whether or not the sample will be excluded. This population will be used for reporting of PK data. |
| Hypothesis | This study is designed to estimate the relative BA of each test treatment to the reference treatment (B vs. A, C vs. A in Part 1; E vs. D, F vs. D in Part 2) in the fasted state. |
| | <ul> <li>No formal hypothesis will be tested. For each primary pharmacokinetic endpoint (AUC[0-∞], AUC[0-t], and Cmax), point estimates and corresponding 90% CIs will be constructed for the ratio of the geometric mean of the test treatment to the geometric mean of the reference treatment, µ(test)/µ(reference).</li> </ul> |

### 2. SUMMARY OF KEY PROTOCOL INFORMATION

### 2.1. Changes to the Protocol Defined Statistical Analysis Plan

An additional comparison between the two administration approaches of Pediatric TRIUMEQ in Part 1 and Pediatric DTG/3TC in Part 2, direct to mouth and dispersion (B vs. C, and E vs. F) will be included within the primary statistical analyses. The secondary PK parameter C24 will be included in the primary statistical analysis described in Section 7.1.3.2 of this document.

Screened and Enrolled populations have been defined as additional analysis populations.

There have been no other changes to the protocol defined statistical analysis plan.

# 2.2. Study Objective(s) and Endpoint(s)

| Objectives | Endpoints |
|---|---|
| Primary Objectives | Primary Endpoints |
| Part 1 | Part 1 |
| To compare the relative BA of DTG, ABC, and 3TC administered as pediatric TRIUMEQ dispersible tablets with the conventional adult TRIUMEQ tablet (reference) administered as direct-to-mouth when: Pediatric TRIUMEQ dispersible tablets are administered as a dispersion and taken immediately Pediatric TRIUMEQ dispersible tablets are administered as direct to-mouth | <ul> <li>Plasma DTG, ABC, and 3TC:</li> <li>AUC(0-∞), AUC(0-t), and Cmax.</li> </ul> |
| Part 2 | Part 2 |
| To compare the relative BA of DTG and 3TC administered as pediatric DTG/3TC dispersible tablets with the conventional adult DTG and 3TC tablets (reference) administered as direct-to-mouth when: Pediatric DTG/3TC dispersible tablets are administered as a dispersion and taken immediately Pediatric DTG/3TC dispersible tablets are administered as direct-to-mouth | <ul> <li>Plasma DTG and 3TC:</li> <li>AUC(0-∞), AUC(0-t), and Cmax.</li> </ul> |

| Objectives | Fuelmainte |
|---|---|
| Objectives | Endpoints Secondary Endpoints |
| Secondary Objectives | Secondary Endpoints |
| <ul> <li>Part 1</li> <li>To compare the single-dose pharmacokinetics (PK) of DTG, ABC, and 3TC administered as pediatric TRIUMEQ dispersible tablets with the conventional adult TRIUMEQ tablets (reference) administered as direct-to-mouth when: <ul> <li>Pediatric TRIUMEQ dispersible tablets are administered as a dispersion and taken immediately</li> <li>Pediatric TRIUMEQ dispersible tablets are administered as direct to-mouth</li> </ul> </li> <li>To evaluate the safety and tolerability of DTG, ABC, and 3TC administered as pediatric TRIUMEQ dispersible tablets as compared with conventional adult TRIUMEQ tablet (reference) administered as direct-to-mouth.</li> </ul> | <ul> <li>Part 1</li> <li>Plasma DTG, ABC, and 3TC: AUC(0-24), Tmax, Tlast, CL/F, Vz/F, C24, Ct, t½</li> <li>Plasma DTG: tlag</li> <li>Safety and tolerability parameters for AEs/SAEs, observed and change from baseline clinical laboratory assessments, ECG, and vital signs.</li> </ul> |
| <ul> <li>To compare the single-dose pharmacokinetics (PK) of DTG and 3TC administered as pediatric DTG/3TC dispersible tablets, with the conventional adult DTG and 3TC tablets (reference) administered as direct-to-mouth when: <ul> <li>Pediatric DTG/3TC dispersible tablets are administered as a dispersion and taken immediately</li> <li>Pediatric DTG/3TC dispersible tablets are administered as direct to-mouth</li> </ul> </li> <li>To evaluate the safety and tolerability of DTG and 3TC administered as pediatric DTG/3TC dispersible tablets as compared with the conventional adult DTG and 3TC tablets (reference) administered as direct-to-mouth</li> </ul> | <ul> <li>Part 2</li> <li>Plasma DTG and 3TC: AUC(0-24), Tmax, Tlast, CL/F, Vz/F, C24, Ct, t½</li> <li>Plasma DTG: tlag</li> <li>Safety and tolerability parameters for AEs/SAEs, observed and change from baseline clinical laboratory assessments, ECG, and vital signs.</li> </ul> |
| Exploratory Objectives | Exploratory Endpoints |
| Parts 1 and 2 | Parts 1 and 2 |
| To evaluate the palatability of the dispersible tablets. | Palatability questionnaire. |

### 2.3. Study Design



| Overview of Study Des | ign and Key Features |
|---|---|
| | <ul> <li>Part 2:</li> <li>Treatment D: Adult DTG (50 mg, 1 conventional tablet) and adult 3TC (300 mg, 1 conventional tablet) administered as direct-to-mouth (reference)</li> <li>Treatment E: Pediatric DTG/3TC (DTG 5 mg/3TC 30 mg, 10 dispersible tablets) administered as a dispersion and taken immediately (test).</li> <li>Treatment F: Pediatric DTG/3TC (DTG 5 mg/3TC 30 mg, 10 dispersible tablets) administered as direct-to-mouth (test).</li> </ul> |
| Treatment<br>Assignment | <ul> <li>Part 1:</li> <li>On Period 1 Day 1, participants will be randomized to 1 of the 6 following treatment sequences: ABC, BCA, CAB, ACB, BAC, or CBA in accordance with the randomization schedule generated prior to the start of the study, using validated software.</li> <li>Part 2:</li> <li>On Period 1 Day 1, participants will be randomized to 1 of the 6 following treatment sequences: DEF, EFD, FDE, DFE, EDF, or FED in accordance with the randomization schedule generated prior to the start of the study, using validated software.</li> </ul> |
| Interim Analysis | There will be no interim analysis. |

### 2.4. Statistical Hypotheses

This study is designed to estimate the relative BA of each test treatment to the reference treatment (B vs. A, C vs. A; E vs. D, F vs. D) in both study parts in the fasted state. Administration by either direct to mouth or dispersion will also be directly compared (B vs. C, and E vs. F) in both study parts.

No formal hypothesis will be tested. For each primary pharmacokinetic endpoint  $(AUC[0-\infty], AUC[0-t], and Cmax)$ , point estimates and corresponding 90% CIs will be constructed for the ratio of the geometric mean of the test treatment to the geometric mean of the reference treatment,  $\mu(test)/\mu(reference)$ .

### 3. PLANNED ANALYSES

### 3.1. Final Analyses

The final planned primary analyses will be performed after the completion of the following sequential steps:

- 1. All participants have completed the study as defined in the protocol
- 2. All required database cleaning activities have been completed and final database release and database freeze has been declared by Data Management.

### 4. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| Screened | All participants who signed an informed | <ul> <li>Screen Failures</li> </ul> |
| | consent form. | <ul> <li>Protocol Deviations</li> </ul> |
| Enrolled | All participants who were randomized | <ul> <li>Study Populations</li> </ul> |
| All Participants | All participants who receive at least one dose | <ul> <li>Demographic</li> </ul> |
| | of study medication. This population | <ul> <li>Safety</li> </ul> |
| | corresponds to all participants enrolled. | <ul> <li>Exploratory</li> </ul> |
| PK | Participants in the "All Participants" population for whom a PK sample was obtained and who had evaluable PK assay results. PK samples that may be affected by protocol deviations will be reviewed by the study team to determine whether or not the sample will be excluded. | • PK |

#### NOTES:

 Please refer to Appendix 10: List of Data Displays which details the population to be used for each display being generated.

### 4.1. Protocol Deviations

- Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be summarised and listed.
- Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan.
  - Data will be reviewed prior to freezing the database to ensure all important deviations and deviations which may lead to exclusion from the analysis are captured and categorised on the protocol deviations dataset.
  - This dataset will be the basis for the summaries and listings of protocol deviations.
- A separate summary and listing of all inclusion/exclusion criteria deviations will also be provided. This summary will be based on data as recorded on the inclusion/exclusion page of the electronic case report form (eCRF).

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

Table 1 provides an overview of appendices within the RAP for outlining general considerations for data analyses and data handling conventions.

Table 1 Overview of Appendices

| Section | Component |
|---|---|
| 10.1 | Appendix 1: Time & Events |
| 10.2 | Appendix 2: Treatment States and Phases |
| 10.3 | Appendix 3: Data Display Standards & Handling Conventions |
| 10.4 | Appendix 4: Derived and Transformed Data |
| 10.5 | Appendix 5: Premature Withdrawals & Handling of Missing Data |
| 10.6 | Appendix 6: Values of Potential Clinical Importance |
| 10.7 | Appendix 7: Multiple Comparisons and Multiplicity |
| 10.8 | Appendix 8: Model Checking and Diagnostics for Statistical Analyses. |
| 10.9 | Appendix 9: Abbreviations and Trade Marks |
| 10.10 | Appendix 10: List of Data Displays |
| 10.11 | Appendix 11: Example Mock Shells for Data Displays |

### 6. STUDY POPULATION ANALYSES

# 6.1. Overview of Planned Analyses

The study population analyses will be based on the "All Participants" population, unless otherwise specified.

Table 2 provides an overview of the planned study population analyses, with full details of data displays being presented in Appendix 10: List of Data Displays.

 Table 2
 Overview of Planned Study Population Analyses

| Display Type | Data Display | Data Display's Generated | |
|---|---|---|---|
| | Figure | Table | Listing |
| Enrollment | | | |
| Number of Participants Enrolled by Country and Site ID | | Υ | |
| Randomisation | • | | |
| Randomisation | | | Υ |
| Participant Disposition | | | |
| Participant Disposition | | Y | |
| Reasons for Screen Failures | | Y | Υ |
| Reasons for Withdrawals | | | Υ |
| Important Protocol Deviations | | Υ | Υ |
| Inclusion and Exclusion Criteria Deviations | | | Υ |
| Demography | | | |
| Demographics Characteristics | | Y | Υ |
| Race and Racial Combinations | | Y | Υ |
| Age Ranges | | Y | |
| Study Populations | | | Υ [1] |
| Concomitant Medications | | | |
| Concomitant Medications | | | Υ |

#### NOTES:

- Y = Yes display generated.
- 1. Listing includes only participants excluded from any population.

### 7. PRIMARY STATISTICAL ANALYSES

### 7.1. Pharmacokinetic Analyses

### 7.1.1. Overview of Planned Pharmacokinetic Analyses

The PK analyses will be based on the PK Population, unless otherwise specified.

Table 3 provides an overview of the planned analyses, with full details being presented in Appendix 10: List of Data Displays.

Table 3 Overview of Planned Pharmacokinetic Analyses

| Display Type | Untransformed | | | | | | Ln-Transformed | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Stats Analysis | | ysis Summary | | Individual | | Stats Analysis | | ysis | Summary | | Individual | | |
| | Т | F | L | T | F | F | L | Т | F | L | Т | F | F | L |
| PK Concentrations | | | | Υ | <b>Y</b> [1] | <b>Y</b> [1] | Y | | | | | | | |
| Plasma PK<br>Parameters | Υ | | | Υ | <b>Y</b> [1] | Υ | Υ | | | Υ | Υ | | | |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual participant observed raw data.
- 1. [1] Linear and Semi-Logarithmic plots will be created on the same display.
- 2. [2] Separate mean and median plots will be generated.

### 7.1.2. Drug Concentration Measures

Refer to Appendix 3: Data Display Standards & Handling Conventions (Section 10.3.3 Reporting Process & Standards).

#### 7.1.3. Pharmacokinetic Parameters

### 7.1.3.1. Deriving Pharmacokinetic Parameters

- Refer to Appendix 3: Data Display Standards & Handling Conventions (Section 10.3.3 Reporting Process & Standards).
- The PK parameters will be calculated by standard non-compartmental analysis according to current working practices and using Phoenix WinNonlin Version 6.4 or higher.
- All calculations of non-compartmental parameters will be based on actual sampling times.
- Pharmacokinetic parameters described in Table 4 will be determined from the plasma concentration-time data, as data permits.

 Table 4
 Derived Plasma Pharmacokinetic Parameters

| Parameter | Parameter Description |
|---|---|
| AUC(0-t) | Area under the concentration-time curve (AUC) from time 0 (predose) to time of the last quantifiable concentration, to be calculated using the linear trapezoidal rule for each incremental trapezoid and the log trapezoidal rule for each decremental trapezoid. |
| AUC(0-24) | Area under the concentration-time curve (AUC) over time 0 (predose) to 24 hours after dose administration, to be calculated using the linear trapezoidal rule for each incremental trapezoid and the log trapezoidal rule for each decremental trapezoid. |
| AUC(0-∞) | Area under the concentration-time curve from time 0 (predose) extrapolated to infinite time, calculated as: |
| | $AUC(0-\infty) = AUC(0-t) + Ct / \lambda z$ |
| | where Ct is the last observed quantifiable concentration. |
| %AUCex | The percentage of AUC(0-∞) obtained by extrapolation (%AUCex) will be calculated as: |
| | [AUC(0-∞) – AUC(0-t)] / AUC(0-∞) x 100 |
| Cmax | Maximum observed concentration, determined directly from the concentration-time data. |
| Ct | The last observed quantifiable concentration |
| C24 | The observed concentration at 24 hours after dose administration |
| Tmax | Time to first occurrence of Cmax |
| Tlast | Time of last quantifiable concentration |
| tlag | Lag time before observation of drug concentrations in sampled matrix |
| t½ | Terminal phase half-life will be calculated as: |
| | $t\frac{1}{2} = \ln 2 / \lambda z$ |
| λz | Terminal-phase rate constant |
| CL/F | The apparent oral clearance |
| Vz/F | The apparent volume of distribution during the terminal phase |

### NOTES:

- Additional parameters may be included as required.
- tlag will be calculated for DTG only

### 7.1.3.2. Statistical Analysis of Pharmacokinetic Parameters

The following PK statistical analyses will only be performed, if sufficient data are available (i.e. if participants have well defined plasma profiles).

### **Pharmacokinetic Statistical Analyses**

### Endpoint(s)

• Plasma primary PK endpoints include AUC(0-∞), AUC(0-t) and Cmax and the secondary endpoint C24 for DTG, ABC (only for Part 1), and 3TC, as data permit

### **Model Specification**

- In Part 1 of this study, the In-transformed AUC(0-∞), AUC(0-t), Cmax, and C24 values for DTG, ABC, and 3TC will be analyzed separately using a mixed effects model, fitting fixed effect terms for period, treatment, and treatment sequence; and treating participant within treatment sequence as a random effect. Point estimates and 90% CIs will be constructed using the residual variance for the following differences of interest:
  - 10 dispersible pediatric TRIUMEQ tablets [DTG 5 mg/ABC 60 mg/3TC 30 mg] administered as a dispersion and taken immediately [Treatment B, Test] and administered direct-to-mouth [Treatment C, Test] versus 1 conventional adult TRIUMEQ tablet [DTG 50 mg/ABC 600 mg/3TC 300 mg] administered direct-tomouth [Treatment A, Reference]
  - 10 dispersible pediatric TRIUMEQ tablets [DTG 5 mg/ABC 60 mg/3TC 30 mg] administered as a dispersion and taken immediately [Treatment B, Test] versus 10 dispersible pediatric TRIUMEQ tablets [DTG 5 mg/ABC 60 mg/3TC 30 mg] administered direct-to-mouth [Treatment C, Reference])
- In Part 2 of this study, the In-transformed AUC(0-∞), AUC(0-t), Cmax, and C24 values for DTG and 3TC will be analyzed separately using a mixed effects model, fitting fixed effect terms for period, treatment, and treatment sequence; and treating participant within treatment sequence as a random effect. Point estimates and 90% CIs will be constructed using the residual variance for the following differences of interest:
  - 10 dispersible pediatric DTG/3TC tablets [DTG 5 mg/3TC 30 mg] administered as a dispersion and taken immediately [Treatment E, Test] and administered directto-mouth [Treatment F, Test] versus 1 conventional adult DTG tablet [50mg] and 1 conventional 3TC tablet [300 mg] administered direct-to-mouth [Treatment D, Reference]
  - 10 dispersible pediatric DTG/3TC tablets [DTG 5 mg/3TC 30 mg] administered as a dispersion and taken immediately [Treatment E, Test] versus 10 dispersible pediatric DTG/3TC tablets [DTG 5 mg/3TC 30 mg] administered direct-to-mouth [Treatment F, Reference])

### **Model Checking & Diagnostics**

Refer to Appendix 8: Model Checking and Diagnostics for Statistical Analyses.

#### **Model Results Presentation**

 Statistical analysis by ANOVA will be presented in tabular format with geometric mean ratios between TRIUMEQ dispersible pediatric tablets versus conventional adult tablets and TIRUMEQ dispersible pediatric tablets administered as a dispersion versus TRIUMEQ dispersible pediatric tablets administered as direct-to-mouth (Part 1) and DTG/3TC dispersible pediatric tablets versus conventional adult tablets and DTG/3TC dispersible pediatric tablets

### **Pharmacokinetic Statistical Analyses**

administered as a dispersion versus DTG/3TC dispersible pediatric tablets administered as direct-to-mouth (Part 2), and 90% CIs for the ratios of AUC( $0-\infty$ ), AUC(0-t), Cmax, and C24 for DTG, ABC (only for Part 1), and 3TC.

Part 1 Example SAS Code:

PROC MIXED;

CLASS USUBJID TRTA TRTSEQP APERIOD;

MODEL LOGPKPARM =TRTA TRTSEQP APERIOD /DDFM=KR;

RANDOM USUBJID(TRTSEQP);

LSMEANS TRTA;

ESTIMATE 'B VS A' TRTA -1 1 0/CL ALPHA=0.1;

ESTIMATE 'C VS A' TRTA -1 0 1/CL ALPHA=0.1;

ESTIMATE 'B VS C' TRTA 0 1-1/CL ALPHA=0.1;

RUN;

Part 2 Example SAS Code:

PROC MIXED;

CLASS USUBJID TRTA TRTSEQP APERIOD;

MODEL LOGPKPARM =TRTA TRTSEQP APERIOD /DDFM=KR;

RANDOM USUBJID(TRTSEQP):

LSMEANS TRTA;

ESTIMATE 'E VS D' TRTA -1 1 0/CL ALPHA=0.1;

ESTIMATE 'F VS D' TRTA -1 0 1/CL ALPHA=0.1;

ESTIMATE 'E VS F' TRTA 0 1-1/CL ALPHA=0.1;

RUN;

### 7.1.4. Interim Analysis

### 7.1.4.1. Overview of Planned Analyses

No interim analysis is planned for this study.

# 8. SECONDARY STATISTICAL ANALYSES

# 8.1. Safety Analyses

The safety analyses will be based on the "All Participants" population, unless otherwise specified.

Table 5 provides an overview of the planned analyses, with further details of data displays being presented in Appendix 10: List of Data Displays.

Table 5 Overview of Planned Safety Analyses

| Display Type | Absolute | | | ( | Change from Baseline | | | |
|---|---|---|---|---|---|---|---|---|
| | Sur | nmary | Indiv | ridual | Sum | mary | Indiv | ridual |
| | Т | F | F | L | Т | F | F | L |
| Exposure | | | | | | | | |
| Exposure Data | | | | Υ | | | | |
| Adverse Events | | | | | | | | |
| Relationship Between | | | | Υ | | | | |
| System Organ Class and | | | | | | | | |
| Verbatim Term | | | | | | | | |
| Subject Numbers for | | | | Υ | | | | |
| Individual AEs | | | | | | | | |
| All AEs | Υ | | | Υ | | | | |
| All Drug-Related AEs | Υ | | | Υ | | | | |
| Common Non-serious | Y | | | | | | | |
| AEs | | | | | | | | |
| Serious AEs | Υ | | | Υ | | | | |
| AEs by Maximum Grade | Υ | | | | | | | |
| Withdrawal AEs | | | | Υ | | | | |
| Laboratory Values | | | | | | | | |
| Clinical Chemistry | Υ | | | Υ [2] | Υ | | | |
| Hematology | Υ | | | Υ [2] | Υ | | | |
| Urinalysis (Dipstick) | <b>Y</b> [5] | | | Υ [2] | | | | |
| Electrocardiograms (ECG | Ss) | | | | | | | |
| ECG Findings | Υ | | | Y [3] | | | | |
| ECG Values | Υ | | | Y [4] | | | | |
| Vital Signs | | | | | | | | |
| Vital Signs | Υ | | | Y [4] | Υ | | | |
| Liver | | | | | | | | |
| Liver Events [1] | | | | Υ | | | | |

#### NOTES:

- 1. Conditional display, it will only be produced when an event has occurred.
- 2. Displays contain only participants with DAIDS toxicities for HIV-infected patients of Grade 2 or higher
- 3. Displays contain only participants with abnormal findings
- 4. Displays contain only participants with values of potential clinical importance
- 5. Displays contain only worst case results relative to baseline
- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents TFL related to any displays of individual participant observed raw data.

### 8.2. Exploratory Analyses

The exploratory analyses will be based on the "All Participants" population, unless otherwise specified.

Table 6 provides an overview of the planned analyses, with further details of data displays being presented in Appendix 10: List of Data Displays.

Table 6 Overview of Planned Exploratory Analyses

| Display Type | Absolute | | | |
|------------------------------------|----------|------|------------|---|
| | Sum | mary | Individual | |
| | T | F | F | L |
| Palatability | | | | |
| Palatability Questionnaire Results | Y | | | Y |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual participant observed raw data.

# 9. REFERENCES

GlaxoSmithKline Document Number 2017N330422\_00 (Original – 18-JAN-2018): 2-Part, Phase I, Single-Dose, 3-Period Crossover Relative Bioavailability Study of a Pediatric TRIUMEQ Dispersible Tablet and Pediatric Dolutegravir and Lamivudine (DTG/3TC) Fixed Dose Combination Dispersible Tablet Formulations as Compared With Adult Tablets in Healthy Volunteers (18-JAN-2018)

# 10. APPENDICES

| Section | Appendix |
|---|---|
| RAP Section 5 | : General Considerations for Data Analyses & Data Handling Conventions |
| Section 10.1 | Appendix 1: Time and Events |
| Section 10.2 | Appendix 2: Treatment States & Phases |
| Section 10.3 | Appendix 3: Data Display Standards & Handling Conventions |
| | Study Treatment & Sub-group Display Descriptors |
| | Baseline Definitions & Derivations |
| | Reporting Process & Standards |
| Section 10.4 | Appendix 4: Derived and Transformed Data |
| | General, Study Population & Safety |
| | Pharmacokinetic |
| | Exploratory |
| Section 10.5 | Appendix 5: Premature Withdrawals & Handling of Missing Data |
| | Premature Withdrawals |
| | Handling of Missing Data |
| Section 10.6 | Appendix 6: Values of Potential Clinical Importance |
| Section 10.7 | Appendix 7: Multiple Comparisons and Multiplicity |
| Section 10.8 | Appendix 8: Model Checking and Diagnostics for Statistical Analyses |
| Other RAP App | endices |
| Section 10.9 | Appendix 9: Abbreviations & Trade Marks |
| Section 10.10 | Appendix 10: List of Data Displays |
| Section 10.11 | Appendix 11: Example Mock Shells for Data Displays |

# 10.1. Appendix 1: Time & Events

# 10.1.1. Protocol Defined Screening Assessments for Parts 1 and 2

| Event | Notes |
|---|---|
| Informed Consent | |
| Demographics | |
| Medical History (includes substance use) | |
| Inclusion/Exclusion | |
| Human Immunodeficiency Virus, Hepatitis B and Hepatitis C Screen | |
| HLA-B*5701 | For Part 1 only. |
| Urine Drug/Alcohol/Cotinine Screen | |
| Physical Examination | A brief physical examination is required at Screening. |
| Height, Weight & Body Mass Index | |
| Vital Sign Measurement | |
| 12-lead Electrocardiogram (Single) | A single repeat evaluation is allowed for eligibility determination. |
| Follicle-stimulating Hormone and Estradiol (women) | |
| Pregnancy Test (urine) | For women of child bearing potential (WOCBP) only. |
| Clinical Laboratory Tests (Chemistry, Hematology, and Urinalysis) | For clinical laboratory tests, see Appendix 2 in the protocol. |
| Concomitant Medication | |

# 10.1.2. Protocol Defined Time and Events for Parts 1 and 2

| | Periods 1-3 | | | | | | | | Notes |
|---|---|---|---|---|---|---|---|---|---|
| | | | | Day<br>1 | Day<br>2 | Day<br>3 | Day<br>4 | dn-v | <ul> <li>Day -1 of Periods 2 and 3 may be the same day as Day 6<br/>of prior periods.</li> </ul> |
| Assessments | Day<br>−1 | Predose | 0<br>hr | Postdose | 24<br>hr | 48<br>hr | 72<br>hr | Follow-up | <ul> <li>At Follow-up, male participants and female participants of<br/>non-childbearing potential with no ongoing AEs or vital<br/>sign/clinical laboratory results of clinical concern may be<br/>followed up virtually by the site via telephone contact.</li> </ul> |
| Admission to Unit | Χ | | | | | | | | |
| Discharge | | | | | | | Х | | |
| Outpatient Visit | | | | | | | | Χ | Follow-up visit will occur 7-10 days after last dose. |
| 12-lead ECG (single) | Χ | | | | | | | | |
| Vital signs | х | Х | | At 4 hours postdose | Х | | | Х | <ul> <li>Single vital sign measurements performed at all time points.</li> <li>Vital signs at Follow-up are only necessary if participant had ongoing AEs or a previous abnormal vital sign result of clinical concern. Only the abnormal value(s) need be re-assessed.</li> </ul> |
| Brief Physical Examination | Х | | | | | | | | Physical examination required only on Day −1 of Period 1 and as needed based on AE assessment. |
| Urine Drug/Alcohol/Cotinine | Χ | | | | | | | | Drug/Alcohol/Cotinine/pregnancy will be performed as per the |
| Pregnancy test (serum; WOCBP) | Χ | | | | | | | Χ | standard practice of the site. |
| Clinical laboratory tests | Х | | | | Х | | | Х | <ul> <li>For clinical laboratory tests, see Appendix 2 in the protocol.</li> <li>Clinical laboratory tests at Follow-up are only necessary if participant had ongoing AEs or a previous abnormal clinical laboratory result of clinical concern. Only the abnormal value(s) need be re-assessed.</li> </ul> |
| Dosing | | | X | | | | | | Participants in Part 1 should be provided with an ABC HSR warning card and should be reminded to read it. |
| Palatability Assessment | | | | Start within 10 minutes after dose | | | | | Complete for each dispersion treatment (Treatments B & E, see Appendix 4 in the protocol). |
| Pharmacokinetic Sampling | | Х | | Collect at: 0.25, 0.5, 1, 8, 12, 16, 24, 48 and before discharge at the | 72 hou | rs postd | lose | | Predose is within 15 minutes prior to dosing (see Section 9.5.1 in the protocol). |

| | Periods 1-3 | | | | | | | Notes | |
|---|---|---|---|---|---|---|---|---|---|
| | Day<br>−1 | Day<br>1 | | | Day<br>2 | Day<br>3 | Day<br>4 | dn-v | |
| Assessments | | Predose | 0<br>hr | Postdose | 24<br>hr | 48<br>hr | 72<br>hr | Follow | At Follow-up, male participants and female participants of<br>non-childbearing potential with no ongoing AEs or vital<br>sign/clinical laboratory results of clinical concern may be<br>followed up virtually by the site via telephone contact. |
| Meals | | ed from 10 h<br>o dosing to 4<br>postdos | hours | r<br>Standard for | the stud | y centre | | | |
| Adverse Events / SAE | Χ | <b>←</b> ===== | | =====X====== | ===== | | == <b>→</b> | Χ | |
| Concomitant medications | Χ | <b>←</b> | | | <del>-</del> | Χ | | | |

# 10.2. Appendix 2: Treatment States and Phases

### 10.2.1. Treatment States

Assessments and events will be classified according to time of occurrence relative to the start and/or stop date of the study treatment.

### 10.2.1.1. Treatment States for Safety Data

| Treatment State | Definition |
|---|---|
| Pre-Treatment | Date/Time < Study Treatment Start Date/Time |
| On-Treatment | Study Treatment Start Date/Time ≤ Date/Time ≤ Study Treatment Stop Date/Time + 6 days |
| Post-Treatment | Date/Time > Study Treatment Stop Date/Time + 6 days |

### 1. NOTES:

• If the study treatment stop date is missing then the assessment will be considered to be On-Treatment

### 10.2.1.2. Treatment States for Event Data (e.g. AEs, Concomitant Medications)

| Treatment State | Definition |
|---|---|
| Pre-Treatment | Event Start Date/Time < Initial Study Treatment Date/Time |
| On-Treatment | If event onset date/time is on or after the initial treatment date/time & on or before the final treatment date/time with 7 days lag time. Initial Study Treatment Date/Time ≤ Event Start Date/Time ≤ Final Study Treatment Date/Time + 6 days |
| Post-Treatment | If event onset date/time is after the final treatment date/time with 6 days lag time. Event Start Date/Time > Final Study Treatment Date/Time + 6 days |
| Onset Time<br>Since 1st Dose<br>(Days) | If Treatment Date/Time > Event Onset Date/Time = Event Onset Date – Treatment Date/Time If Treatment Date/Time ≤ Event Onset Date/Time = Event Onset Date/Time – Treatment Date/Time +1 Missing otherwise. |
| Duration (Days) | Event Resolution Date/Time – Event Onset Date/Time + 1 |
| Drug-related | If relationship is marked 'YES' on eCRF OR value is missing. |

#### NOTES:

• If the initial and final study treatment dates are missing then the event will be considered to be On-Treatment.

# 10.3. Appendix 3: Data Display Standards & Handling Conventions

### 10.3.1. Study Treatment & Sub-group Display Descriptors

| | Treatment Group Descriptions | | | |
|---|---|---|---|---|
| Study | | Treatment Group | Data Displays for Reporting | |
| Part | Code | Description | Description <sup>[1]</sup> | Order [2] |
| 1 | Α | Adult TRIUMEQ (DTG 50 mg/ABC 600 mg/3TC 300 mg, 1 conventional tablet) administered as direct-to-mouth (reference) | Treatment A | 1 |
| | В | Pediatric TRIUMEQ (DTG<br>5 mg/ABC 60 mg/3TC 30 mg,<br>10 dispersible tablets) administered<br>as a dispersion and taken<br>immediately (test) | Treatment B | 2 |
| | С | Pediatric TRIUMEQ (DTG<br>5 mg/ABC 60 mg/3TC 30 mg,<br>10 dispersible tablets) administered<br>as direct-to-mouth (test) | Treatment C | 3 |
| 2 | D | Adult DTG (50 mg, 1 conventional tablet) and adult 3TC (300 mg, 1 conventional tablet) administered as direct-to-mouth (reference) | Treatment D | 4 |
| | E | Pediatric DTG/3TC (DTG<br>5 mg/3TC 30 mg, 10 dispersible<br>tablets) administered as a<br>dispersion and taken immediately<br>(test) | Treatment E | 5 |
| | F | Pediatric DTG/3TC (DTG<br>5 mg/3TC 30 mg, 10 dispersible<br>tablets) administered as direct-to-<br>mouth (test) | Treatment F | 6 |

#### NOTES:

- 1. The word "Treatment" may be omitted from displays in order to limit wrapping
- 2. Order represents treatments being presented in TFL, as appropriate.
- Where applicable, outputs will include a treatment footnote describing the treatments: "Treatment A = Adult TRIUMEQ (DTG 50 mg/ABC 600 mg/3TC 300 mg, 1 conventional tablet) administered as direct-to-mouth (reference); Treatment B = Pediatric TRIUMEQ (DTG 5 mg/ABC 60 mg/3TC 30 mg, 10 dispersible tablets) administered as a dispersion and taken immediately (test); Treatment C = Pediatric TRIUMEQ (DTG 5 mg/ABC 60 mg/3TC 30 mg, 10 dispersible tablets) administered as direct-to-mouth (test); Treatment D = Adult DTG (50 mg, 1 conventional tablet) and adult 3TC (300 mg, 1 conventional tablet) administered as direct-to-mouth (reference); Treatment E = Pediatric DTG/3TC (DTG 5 mg/3TC 30 mg, 10 dispersible tablets) administered as a dispersion and taken immediately (test); Treatment F = Pediatric DTG/3TC (DTG 5 mg/3TC 30 mg, 10 dispersible tablets) administered as direct-to-mouth (test)."

#### 10.3.2. Baseline Definition & Derivations

#### 10.3.2.1. Baseline Definitions

For all endpoints (except as noted in baseline definitions) the baseline value will be the last available assessment prior to time of the first dose, unless noted otherwise. Baseline definitions are applicable to each period. For later periods, Day -1 may be the same day as Day 6 of the prior period.

| Parameter | Study Assess | Baseline Used in | | |
|---|---|---|---|---|
| | Screening | Screening Day -1 Day 1 (Pre-Dos | | Data Display |
| Safety | | | | |
| Hematology | X | Χ | | Day -1 |
| Clinical Chemistry | Х | Χ | | Day -1 |
| 12-Lead ECG | Х | Х | | Day -1 |
| Vital Signs | Х | Χ | Х | Day 1 (Pre-Dose) |

#### NOTES:

• Unless otherwise stated, the mean of replicate assessments at any given time point will be used as the value for that time point.

### 10.3.2.2. Derivations and Handling of Missing Baseline Data

| Definition | Reporting Details |
|----------------------|------------------------------------|
| Change from Baseline | = Post-Dose Visit Value – Baseline |

#### NOTES:

- Unless otherwise specified, the baseline definitions specified in Section 10.3.2.1 Baseline Definitions will be used for derivations for endpoints / parameters and indicated on summaries and listings.
- Unless otherwise stated, if baseline data is missing no derivation will be performed and will be set to missing.
- The baseline definition will be footnoted on all change from baseline displays.

### 10.3.3. Reporting Process & Standards

### Reporting Process

### **Software**

 The currently supported versions of SAS 9.3 or higher and Phoenix WinNonlin software 6.4 or higher will be used.

#### **Analysis Datasets**

- Analysis datasets will be created according to CDISC standards SDTM IG Version 3.2 & ADaM IG Version 1.0.
- For creation of ADaM datasets (ADCM/ADAE), the same version of dictionary datasets will be implemented for conversion from SI to SDTM.

### **Generation of RTF Files**

RTF files will be generated for all reporting efforts described in the RAP.

### **Reporting Standards**

#### General

- The current GSK IDSL will be applied for reporting, unless otherwise stated:
  - 4.03 to 4.23: General Principles
  - 5.01 to 5.08: Principles Related to Data Listings
  - o 6.01 to 6.11: Principles Related to Summary Tables
  - 7.01 to 7.13: Principles Related to Graphics

#### **Formats**

- All data will be reported according to the actual treatment the participant received unless otherwise stated.
- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places will be adopted for reporting
  of data based on the raw data collected.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.

#### Planned and Actual Time

- Reporting for tables, figures and formal statistical analyses:
  - Planned time relative to dosing will be used in figures (with the exception of individual PK concentration-time figures, where actual relative time will be used), summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the participant's listings.
  - Visits outside the protocol defined time-windows (i.e. recorded as protocol deviations) will be included in listings but omitted from figures, summaries and statistical analyses.

### **Unscheduled Visits**

- Unscheduled visits will not be included in summary tables.
- Unscheduled visits will not be included in figures.
- All unscheduled visits will be included in listings.

### **Descriptive Summary Statistics**

### Continuous Data

Refer to IDSL Statistical Principle 6.06.1

- NQs at the beginning of a participant profile (i.e. before the first incidence of a measurable concentration) are deemed to be zero as it is assumed that in this circumstance no drug is yet measurable in the blood.
- For NQs at the end of the participant profile (i.e. after the last incidence of a measurable concentration);
  - for individual plots and pharmacokinetic analyses these are dropped (set to missing) as they do not provide any useful information (and can erroneously indicate that absolutely no drug is present)

| Reporting Standard | S |
|---|---|
| | <ul> <li>for summary statistics these are set to 0 (to avoid skewing of the summary statistics)</li> <li>Individual NQs which fall between two measurable concentrations are set to missing (individual values of this nature are assumed to be an anomaly)</li> <li>If two or more NQ values occur in succession between measurable concentrations, the profile will be deemed to have terminated at the last measurable concentration prior to these NQs. For the purpose of individual participant plots, these NQs will be set to 0, and the subsequent measurable concentrations will be retained. For the derivation of pharmacokinetic parameters, these NQs and any subsequent measurable concentrations will be omitted (set to missing).</li> </ul> |
| Categorical Data | N (number of participants in subgroup), n (number of participants with evaluable data), frequency, % |
| Reporting of Pharm | acokinetic Concentration Data |
| Descriptive<br>Summary Statistics | Refer to IDSL Statistical Principle 6.06.1 Assign zero to NQ values (Refer to GUI_51487 for further details) |
| Reporting of Pharm | acokinetic Parameters |
| Descriptive<br>Summary Statistics<br>(Ln-Transformed) | N (number of participants in subgroup), n (number of participants with evaluable data), geometric mean, 95% CI of geometric mean, standard deviation (SD) of logged data and between geometric coefficient of variation (CVb (%)) will be reported. CV <sub>b</sub> (%) = square root of (exp(SD <sup>2</sup> ) – 1) * 100 (SD = SD of In-transformed data) |
| Parameters Not<br>Being Ln-<br>Transformed | Tmax, Tlast, tlag, first point, last point, and number of points used in the determination of $\lambda z$ , %AUCex. |
| Summary Tables | The following PK parameters will not be summarised: first point, last point, and number of points used in the determination of λz and Rsq_adjusted. |
| Listings | Include the first point, last point and number of points used in the determination of λz. nd Rsq_adjusted for listings |
| <b>Graphical Displays</b> | |
| Refer to IDSL Sta | atistical Principals 7.01 to 7.13. |

### 10.4. Appendix 4: Derived and Transformed Data

#### 10.4.1. General

### **Multiple Measurements at One Time Point**

- Mean of the measurements will be calculated and used in any derivation of summary statistics but if listed, all data will be presented.
- If there are two values within a time window the value closest to the target day for that window will be used. If values are the same distance from the target then the mean will be taken.
- Participants having both High and Low values for Normal Ranges at any post-baseline visits for safety parameters will be counted in both the High and Low categories of "Any visit postbaseline" row of related summary tables. This will also be applicable to relevant Potential Clinical Importance summary tables.

### **Study Day**

- Calculated as the number of days from randomisation date:
  - Ref Date = Missing
- → Study Day = Missing
- Ref Date < Randomisation Date → Study Day = Ref Date Randomisation Date
- Ref Data ≥ Randomisation Date → Study Day = Ref Date (Randomisation Date) + 1

### 10.4.2. Study Population

### **Demographics**

### Age

- GSK standard IDSL algorithms will be used for calculating age where birth date will be imputed as follows:
  - Only the year of birth will be collected. The date and month will be imputed as '30th June'.
- Birth date will be presented in listings as 'YYYY'.

#### Body Mass Index (BMI)

Calculated as Weight (kg) / [Height (m)<sup>2</sup>]

### 10.4.3. Safety

### **ECG Parameters**

#### RR Interval

- IF RR interval (msec) is not provided directly, then RR can be derived as:
  - [1] If QTcB is machine read & QTcF is not provided, then:

$$RR = \left[ \left( \frac{QT}{QTcB} \right)^2 \right] * 1000$$

[2] If QTcF is machine read and QTcB is not provided, then:

$$RR = \left[ \left( \frac{QT}{OTcF} \right)^3 \right] * 1000$$

If ECGs are manually read, the RR value preceding the measurement QT interval should be a

### **ECG Parameters**

collected value THEN do not derive.

• Machine read values of RR should not be replaced with derived values.

### **Corrected QT Intervals**

- When not entered directly in the eCRF, corrected QT intervals by Bazett's (QTcB) and Fredericia's (QTcF) formulas will be calculated, in msec, depending on the availability of other measurements.
- IF RR interval (msec) is provided then missing QTcB and/or QTcF will be derived as:

$$QTcB = \frac{QT}{\sqrt{\frac{RR}{1000}}}$$

$$QTcF = \frac{QT}{3\sqrt{\frac{RR}{1000}}}$$

### **Adverse Events**

### **AEs of Special Interest**

No analysis for AEs of Special Interest will be performed

# 10.5. Appendix 5: Premature Withdrawals & Handling of Missing Data

### 10.5.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Participant study completion (i.e. as specified in the protocol) was defined as completing all phases of the study including the follow-up visit.</li> <li>Withdrawn participants may be replaced in the study.</li> <li>All available data from participants who were withdrawn from the study will be listed and all available planned data will be included in summary tables and figures, unless otherwise specified.</li> </ul> |

# 10.5.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument: <ul> <li>These data will be indicated by the use of a "blank" in participant listing displays. Unless all data for a specific visit are missing in which case the data is excluded from the table.</li> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to be missing data and should be displayed as such.</li> </ul> </li> </ul> |
| Outliers | Any participants excluded from the summaries and/or statistical analyses will be documented along with the reason for exclusion in the clinical study report. |

# 10.5.2.1. Handling of Missing Dates

| Element | Reporting Detail |
|---|---|
| General | Partial dates will be displayed as captured in participant listing displays. |
| AEs | <ul> <li>The eCRF allows for the possibility of partial dates (i.e., only month and year) to be recorded for AE start and end dates; that is, the day of the month may be missing. In such a case, the following conventions will be applied for calculating the time to onset and the duration of the event: <ul> <li>Missing Start Day: First of the month will be used unless this is before the start date of study treatment; in this case the study treatment start date will be used and hence the event is considered On-treatment as per Appendix 2: Treatment States and Phases.</li> <li>Missing Stop Day: Last day of the month will be used, unless this is after the stop date of study treatment; in this case the study treatment stop date will be used.</li> </ul> </li> <li>Completely missing start or end dates will remain missing, with no imputation applied. Consequently, time to onset and duration of such events will be missing.</li> </ul> |

| Element | Reporting Detail |
|---|---|
| | Start or end dates which are completely missing (i.e. no year specified) will |
| | remain missing, with no imputation applied. |

# 10.5.2.2. Handling of Partial Dates

| Element | Reporting Detail |
|---|---|
| Concomitant<br>Medications | <ul> <li>Partial dates for any concomitant medications recorded in the eCRF will be imputed using the following convention:</li> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month</li> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month.</li> <li>The recorded partial date will be displayed in listings.</li> </ul> |
| AEs | <ul> <li>Any partial dates for AEs will be raised to data management. If the full date cannot be ascertained, the following assumptions will be made: <ul> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month.</li> <li>However, if these results in a date prior to Week 1 Day 1 and the event could possibly have occurred during treatment from the partial information, then the Week 1 Day 1 date will be assumed to be the start date.</li> <li>The AE will then be considered to start on-treatment (worst case).</li> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month.</li> </ul> </li> <li>The recorded partial date will be displayed in listings.</li> </ul> |

#### **Appendix 6: Values of Potential Clinical Importance** 10.6.

#### 10.6.1. **ECG**

| ECG Parameter | Units | Potential Clinically Important Range | |
|---|---|---|---|
| | | Lower | Upper |
| Absolute | | | |
| Absolute QTc Interval | msec | > 450[1] | |
| | | > 450[2] | ≤ 479 <sup>[2]</sup> |
| | | ≥ 480[2] | ≤ 499 <sup>[2]</sup> |
| | | ≥ 500 <sup>[2]</sup> | |
| Absolute PR Interval | msec | < 110[1] | > 220[1] |
| Absolute QRS Interval | msec | < 75[1] | > 110[1] |
| Change from Baseline | | | |
| Increase from Baseline QTc | msec | ≤ 30 <sup>[2]</sup> | |
| | msec | > 30[1] | ≤ 59 <sup>[2]</sup> |
| | msec | ≥ 60 <sup>[2]</sup> | |

### NOTES:

- Represent standard ECG values of PCI for HV studies.
   Represent further subdivisions of ECG values for analysis.

#### 10.6.2. **Vital Signs**

| Vital Sign Parameter | Units | Potential Clinically Important Range | |
|---|---|---|---|
| (Absolute) | | Lower | Upper |
| Systolic Blood Pressure | mmHg | < 85 | > 160 |
| Diastolic Blood Pressure | mmHg | < 45 | > 100 |
| Heart Rate | bpm | < 40 | > 110 |
# 10.7. Appendix 7: Multiple Comparisons & Multiplicity

# 10.7.1. Handling of Multiple Comparisons & Multiplicity

No adjustments for multiplicity will be made.

# 10.8. Appendix 8: Model Checking and Diagnostics for Statistical Analyses

### 10.8.1. Statistical Analysis Assumptions

| Endpoint(s) | <ul> <li>PK endpoints AUC(0-∞), AUC(0-t), Cmax, and C24</li> </ul> |
|---|---|
| Analysis | Mixed Effects |

### **Assumptions:**

- Model assumptions will be applied, but appropriate adjustments may be made based on the data.
- The Kenward and Roger method for approximating the denominator degrees of freedom and correcting for bias in the estimated variance-covariance of the fixed effects will be used.

# 10.9. Appendix 9 – Abbreviations & Trade Marks

### 10.9.1. Abbreviations

| Abbreviation | Description |
|---|---|
| 3TC | Lamivudine |
| ABC | Abacavir |
| ADaM | Analysis Data Model |
| AE | Adverse Event |
| AUC | Area under the concentration-time curve |
| AUC(0-t) | Area under the concentration-time curve from time 0 (predose) to time |
| | of the last quantifiable concentration |
| AUC(0-24) | Area under the concentration-time curve over time 0 (predose) to 24 |
| | hours after dose administration |
| $AUC(0-\infty)$ | Area under the concentration-time curve from time 0 (predose) |
| , | extrapolated to infinite time |
| %AUCex | The percentage of $AUC(0-\infty)$ obtained by extrapolation |
| BA | Bioavailability |
| BMI | Body Mass Index |
| C24 | The observed concentration at 24 hours after dose administration |
| CDISC | Clinical Data Interchange Standards Consortium |
| CL/F | The apparent oral clearance |
| Cmax | Maximum observed concentration |
| CI | Confidence Interval |
| CPK | Creatine phosphokinase |
| Ct | The last observed quantifiable concentration |
| CV | Coefficient of variation |
| $CV_b$ | Coefficient of variation (Between) |
| DAIDS | Division of Acquired Immune Deficiency Syndrome |
| DTG | Dolutegravir |
| ECG | Electrocardiogram |
| eCRF | Electronic Case Report Form |
| GSK | GlaxoSmithKline |
| HSR | Hypersensitivity reaction |
| ICH | International Conference on Harmonisation |
| IDSL | Integrated Data Standards Library |
| kg | Kilograms |
| m | Meters |
| mg | Milligrams |
| msec | Milliseconds |
| PK | Pharmacokinetic |
| QTcF | Fridericia's QT Interval Corrected for Heart Rate |
| QTcB | Bazett's QT Interval Corrected for Heart Rate |
| R&D | Research and Development |
| RAP | Reporting & Analysis Plan |
| SAC | Statistical Analysis Complete |

| Abbreviation | Description |
|---|---|
| SAS | Statistical Analysis Software |
| SD | Standard deviation |
| SDTM | Study Data Tabulation Model |
| TFL | Tables, Figures & Listings |
| t½ | Terminal phase half-life |
| tlag | Lag time before observation of drug concentrations in sampled matrix |
| Tlast | Time of last quantifiable concentration |
| Tmax | Time to first occurrence of Cmax |
| Vz/F | The apparent volume of distribution during the terminal phase |
| λz | terminal phase rate constant |

## 10.9.2. Trademarks

| Trademarks of the GlaxoSmithKline<br>Group of Companies |
|---------------------------------------------------------|
| TRIUMEQ |

| Trademarks not owned by the GlaxoSmithKline Group of Companies |
|----------------------------------------------------------------|
| Phoenix WinNonlin |
| SAS |

# 10.10. Appendix 10: List of Data Displays

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|----------------------------|-------------|-------------|
| Study Population | 1.1 to 1.7 | NA |
| Safety | 2.1 to 2.16 | NA |
| Pharmacokinetic | 3.1 to 3.14 | 3.1 to 3.21 |
| Exploratory (Palatability) | 4.1 | NA |
| Section | List | ings |
| ICH Listings | 1 to 37 | |
| Other (non-ICH) Listings | 38 to 45 | |

### 10.10.1. Mock Example Shell Referencing

Non IDSL specifications will be referenced as indicated.

| Section | Figure | Table | Listing |
|----------------------------|---------|---------|---------|
| Study Population | POP_Fn | POP_Tn | POP_Ln |
| Safety | SAFE_Fn | SAFE_Tn | SAFE_Ln |
| Pharmacokinetic | PK_Fn | PK_Tn | PK_Ln |
| Exploratory (Palatability) | EXP_Fn | EXP_Tn | EXP_Ln |

#### NOTES:

• Non-Standard displays are indicated in the 'IDSL / TST ID / Example Shell' or 'Programming Notes' column as '[Non-Standard] + Reference.'

#### 10.10.2. Deliverable [Priority]

| Delivery [Priority] [1] | Description |
|-------------------------|-------------------------------------|
| SAC [X] | Final Statistical Analysis Complete |

#### NOTES:

1. Indicates priority (i.e. order) in which displays will be generated for the reporting effort.

# 10.10.3. Study Population Tables

| Study P | opulation Tables | s | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Particip | ant Disposition | and Populations | | · | |
| 1.1 | Enrolled | NS1 | Summary of Number of Participants Enrolled by Country and Site ID | | SAC [1] |
| 1.2 | All<br>Participants | ES1A | Summary of Participant Disposition for the Participant Conclusion Record | | SAC [1] |
| 1.3 | Screened | ES6 | Summary of Screening Status and Reasons for Screen Failures | | SAC [1] |
| 1.4 | Screened | DV1 | Summary of Important Protocol Deviations | | SAC [1] |
| Demog | raphics | | | • | |
| 1.5 | All<br>Participants | DM3 | Summary of Demographic Characteristics | | SAC [1] |
| 1.6 | All<br>Participants | DM5 | Summary of Race and Racial Combinations | | SAC [1] |
| 1.7 | All<br>Participants | DM11 | Summary of Age Ranges | | SAC[1] |

# 10.10.4. Safety Tables

| Safety : | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Adverse | e Events | | | | |
| 2.1 | All<br>Participants | AE1CP | Summary of All Adverse Events by System Organ Class and Preferred Term | | SAC [1] |
| 2.2 | All<br>Participants | AE1CP | Summary of Drug-Related Adverse Events | | SAC [1] |
| 2.3 | All<br>Participants | AE15 | Summary of Common (>=5%) Non-serious Adverse Events by System Organ Class and Preferred Term (Number of Participants and Occurrences) | | SAC [1] |
| 2.4 | All<br>Participants | AE16 | Summary of Serious Adverse Events by System Organ Class and Preferred Term (Number of Participants and Occurrences) | | SAC[1] |
| 2.5 | All<br>Participants | AE5A | Summary of Adverse Events by Maximum Grade by System Organ Class and Preferred Term | | SAC [1] |
| Laborat | tory Values | | | | |
| 2.6 | All<br>Participants | LB1 | Summary of Clinical Chemistry Values | | SAC [1] |
| 2.7 | All<br>Participants | LB1 | Summary of Clinical Chemistry Values Change from Baseline | | SAC [1] |
| 2.8 | All<br>Participants | BL | Summary of Clinical Chemistry Results by Maximum Grade Increase Post-Baseline Relative to Baseline | | SAC [1] |
| 2.9 | All<br>Participants | LB1 | Summary of Hematology Values | | SAC [1] |
| 2.10 | All<br>Participants | LB1 | Summary of Hamatology Values Change from Baseline | | SAC [1] |
| 2.11 | All<br>Participants | LB16 | Summary of Hematology Results by Maximum Grade Increase Post-<br>Baseline Relative to Baseline | | SAC [1] |

| Safety : | Safety : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.12 | All<br>Participants | UR1 | Summary of Worst Case Urinalysis Results Post-Baseline Relative to Baseline | | SAC [1] |
| Electrod | ardiograms | | | | |
| 2.13 | All<br>Participants | EG1 | Summary of ECG Findings | | SAC [1] |
| 2.14 | All<br>Participants | EG2 | Summary of ECG Values | | SAC [1] |
| Vital Sig | Vital Signs | | | | |
| 2.15 | All<br>Participants | VS1 | Summary of Values in Vital Signs | | SAC[1] |
| 2.16 | All<br>Participants | VS1 | Summary of Change from Baseline in Vital Signs | | SAC[1] |

### 10.10.5. Pharmacokinetic Tables

| Pharma | Pharmacokinetic : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| PK Con | centration Data | | | | |
| 3.1 | PK | PKCT1 | Summary of DTG Plasma Pharmacokinetic Concentration-Time Data by Study Part and Treatment | | SAC [1] |
| 3.2 | PK | PKCT1 | Summary of ABC Plasma Pharmacokinetic Concentration-Time Data by Treatment | Part 1 only | SAC [1] |
| 3.3 | PK | PKCT1 | Summary of 3TC Plasma Pharmacokinetic Concentration-Time Data by Study Part and Treatment | | SAC [1] |
| PK Deri | ved Parameters | | | | |
| 3.4 | PK | PKPT4 | Summary of Derived DTG Plasma Pharmacokinetic Parameters (Non-Transformed) by Study Part and Treatment | Parameters with units | SAC [1] |
| 3.5 | PK | PKPT4 | Summary of Derived DTG Plasma Pharmacokinetic Parameters (Ln-Transformed) by Study Part and Treatment | Parameters with units | SAC [1] |
| 3.6 | PK | PKPT4 | Summary of Derived ABC Plasma Pharmacokinetic Parameters (Non-Transformed) by Treatment | Parameters with units; Part 1 only | SAC [1] |
| 3.7 | PK | PKPT4 | Summary of Derived ABC Plasma Pharmacokinetic Parameters (Ln-<br>Transformed) by Treatment | Parameters with units; Part 1 only | SAC [1] |
| 3.8 | PK | PKPT4 | Summary of Derived 3TC Plasma Pharmacokinetic Parameters (Non-Transformed) by Study Part and Treatment | Parameters with units | SAC [1] |
| 3.9 | PK | PKPT4 | Summary of Derived 3TC Plasma Pharmacokinetic Parameters (Ln-<br>Transformed) by Study Part and Treatment | Parameters with units | SAC [1] |

| Pharma | Pharmacokinetic : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| PK Anal | ysis Tables | | | | |
| 3.10 | PK | PKPT3 | Statistical Analysis of DTG Plasma Pharmacokinetic Parameters, Study Part 1 | AUC(0-t), AUC(0-∞), Cmax and C24 only by Treatment. Part 1 only. | SAC [1] |
| 3.11 | PK | PKPT3 | Statistical Analysis of DTG Plasma Pharmacokinetic Parameters, Study Part 2 | AUC(0-t), AUC(0-∞), Cmax and C24 only by Treatment. Part 2 only. | SAC [1] |
| 3.12 | PK | PKPT3 | Statistical Analysis of ABC Plasma Pharmacokinetic Parameters, Study Part 1 | AUC(0-t), AUC(0-∞), Cmax and C24 only by Treatment. Part 1 only. | SAC [1] |
| 3.13 | PK | PKPT3 | Statistical Analysis of 3TC Plasma Pharmacokinetic Parameters,<br>Study Part 1 | AUC(0-t), AUC(0-∞), Cmax and C24only by Treatment. Part 1 only. | SAC [1] |
| 3.14 | PK | PKPT3 | Statistical Analysis of 3TC Plasma Pharmacokinetic Parameters,<br>Study Part 2 | AUC(0-t), AUC(0-∞), Cmax and C24only by Treatment. Part 2 only. | SAC [1] |

# 10.10.6. Pharmacokinetic Figures

| Pharma | cokinetic : Figur | es | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Individu | ual Concentration | n Plots | | | , |
| 3.1 | PK | PKCF1X | Individual DTG Plasma Concentration-Time Plots by Participant (Linear and Semi-Logarithmic) | Paginate by Participant | SAC [1] |
| 3.2 | PK | PKCF1X | Individual ABC Plasma Concentration-Time Plots by Participant (Linear and Semi-Logarithmic) | Paginate by Participant; Part 1 only | SAC [1] |
| 3.3 | PK | PKCF1X | Individual 3TC Plasma Concentration-Time Plots by Participant (Linear and Semi-Logarithmic) | Paginate by Participant | SAC [1] |
| Mean / | Median Concent | ration Plots | | | |
| 3.4 | PK | PKCF2 | Mean DTG Plasma Concentration-Time Plots by Treatment (Linear and Semi-Logarithmic) | All treatments for each Part on one page | SAC [1] |
| 3.5 | PK | PKCF2 | Median DTG Plasma Concentration-Time Plots by Treatment (Linear and Semi-Logarithmic) | All treatments for each Part on one page | SAC [1] |
| 3.6 | PK | PKCF2 | Mean ABC Plasma Concentration-Time Plots by Treatment (Linear and Semi-Logarithmic) | All treatments for Part 1 on one page | SAC [1] |
| 3.7 | PK | PKCF3 | Median ABC Plasma Concentration-Time Plots by Treatment (Linear and Semi-Logarithmic) | All treatments for Part 1 on one page | SAC [1] |
| 3.8 | PK | PKCF3 | Mean 3TC Plasma Concentration-Time Plots by Treatment (Linear and Semi-Logarithmic) | All treatments for each Part on one page | SAC [1] |
| 3.9 | PK | PKCF3 | Median 3TC Plasma Concentration-Time Plots by Treatment (Linear and Semi-Logarithmic) | All treatments for each Part on one page | SAC [1] |

| Pharma | Pharmacokinetic : Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| PK Ana | ysis Plots | | | | |
| 3.10 | PK | PKPF3 | Comparative Plot of Individual DTG Plasma Cmax by Treatment (Linear and Semi-Logarithmic) | All treatments for each Part on one page | SAC [1] |
| 3.11 | PK | PKPF3 | Comparative Plot of Individual DTG Plasma AUC(0-t) by Treatment (Linear and Semi-Logarithmic) | All treatments for each Part on one page | SAC [1] |
| 3.12 | PK | PKPF3 | Comparative Plot of Individual DTG Plasma AUC(0-∞) by Treatment (Linear and Semi-Logarithmic) | All treatments for each Part on one page | SAC [1] |
| 3.13 | PK | PKPF3 | Comparative Plot of Individual DTG Plasma C24 by Treatment (Linear and Semi-Logarithmic) | All treatments for each Part on one page | SAC [1] |
| 3.14 | PK | PKPF3 | Comparative Plot of Individual ABC Plasma Cmax by Treatment (Linear and Semi-Logarithmic) | All treatments for Part 1 on one page | SAC [1] |
| 3.15 | PK | PKPF3 | Comparative Plot of Individual ABC Plasma AUC(0-t) by Treatment (Linear and Semi-Logarithmic) | All treatments for Part 1 on one page | SAC [1] |
| 3.16 | PK | PKPF3 | Comparative Plot of Individual ABC Plasma AUC(0-∞) by Treatment (Linear and Semi-Logarithmic) | All treatments for Part 1 on one page | SAC [1] |
| 3.17 | PK | PKPF3 | Comparative Plot of Individual ABC Plasma C24 by Treatment (Linear and Semi-Logarithmic) | All treatments for Part 1 on one page | SAC [1] |
| 3.18 | PK | PKPF3 | Comparative Plot of Individual 3TC Plasma Cmax by Treatment (Linear and Semi-Logarithmic) | All treatments for each Part on one page | SAC [1] |
| 3.19 | PK | PKPF3 | Comparative Plot of Individual 3TC Plasma AUC(0-t) by Treatment (Linear and Semi-Logarithmic) | All treatments for each Part on one page | SAC [1] |
| 3.20 | PK | PKPF3 | Comparative Plot of Individual 3TC Plasma AUC(0-∞) by Treatment (Linear and Semi-Logarithmic) | All treatments for each Part on one page | SAC [1] |
| 3.21 | PK | PKPF3 | Comparative Plot of Individual 3TC Plasma C24 by Treatment (Linear and Semi-Logarithmic) | All treatments for each Part on one page | SAC [1] |

# 10.10.7. Exploratory Tables

| Explora | Exploratory : Tables | | | |
|---|---|---|---|---|
| No. | No. Population IDSL / TST ID / Example Shell Title Programming Notes Deliverable [Priority] | | | |
| Palatabi | Palatability | | | |
| 4.1 | All<br>Participants | EXP_T1 | Summary of Palatability Questionnaire Results (Part 1, Treatment B and Part 2, Treatment E Only) | SAC[1] |

# 10.10.8. ICH Listings

| ICH : Lis | ICH : Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Random | nisation | | | | |
| 1 | All<br>Participants | CP_TA2 | Listing of Randomized and Actual Treatment | | SAC [1] |
| Particip | ant Disposition | | | | |
| 2 | All<br>Participants | ES3 | Listing of Reasons for Study Withdrawal | | SAC [1] |
| 3 | Screened | ES7 | Listing of Reasons for Screen Failure | | SAC [1] |
| 4 | Screened | DV2A | Listing of Important Protocol Deviations | | SAC [1] |
| 5 | All<br>Participants | IE4 | Listing of Participants with Inclusion/Exclusion Criteria Deviations | | SAC[1] |
| 6 | Enrolled | SP3 | Listing of Participants Excluded from Any Population | | SAC [1] |
| 7 | Enrolled | SAFE_L4 | Listing of Participants in Previous Clinical Trial | | SAC [1] |

| ICH : Lis | ICH : Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Demog | raphics | | | | |
| 8 | All<br>Participants | DM4 | Listing of Demographic Characteristics | | SAC [1] |
| 9 | All<br>Participants | DM10 | Listing of Race | | SAC [1] |
| Concon | nitant Medication | ns | | | |
| 10 | All<br>Participants | CM4 | Listing of Concomitant Medications | | SAC[1] |
| Exposu | re | | | | |
| 11 | All<br>Participants | SAFE_L1 | Listing of Exposure Data | | SAC[1] |
| Adverse | e Events | | | | |
| 12 | All<br>Participants | AE2 | Listing of Relationship Between System Organ Class and Verbatim Text | | SAC[1] |
| 13 | All<br>Participants | AE7 | Listing of Subject Numbers for Individual Adverse Events | | SAC[1] |
| 14 | All<br>Participants | AE9CP | Listing of All Adverse Events | | SAC[1] |
| 15 | All<br>Participants | AE9CP | Listing of Study Drug Related Adverse Events | | SAC[1] |
| 16 | All<br>Participants | SAFE_L2 | Listing of Serious Adverse Events | | SAC[1] |
| 17 | All<br>Participants | AE9CP | Listing of Adverse Events Leading to Permanent Discontinuation of Study Treatment or Withdrawal from Study | | SAC[1] |
| 18 | All<br>Participants | SAFE_L3 | Listing of Liver Adverse Events | | SAC[1] |

| ICH : Lis | ICH : Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 19 | All<br>Participants | AE14 | Listing of Reasons for Considering as a Serious Adverse Event | | SAC[1] |
| Laborat | ory Values | | | | |
| 20 | All<br>Participants | LB6 | Listing of Clinical Chemistry Toxicities of Grade 2 or Higher | | SAC [1] |
| 21 | All<br>Participants | LB6 | Listing of All Clinical Chemistry Data for Participants with Toxicities of Grade 2 or Higher | | SAC [1] |
| 22 | All<br>Participants | LB6 | Listing of Hematology Toxicities of Grade 2 or Higher | | SAC [1] |
| 23 | All<br>Participants | LB6 | Listing of All Hematology Data for Participants with Toxicities of Grade 2 or Higher | | SAC [1] |
| 24 | All<br>Participants | LB6 | Listing of Urinalysis Toxicities of Grade 2 or Higher | | SAC [1] |
| 25 | All<br>Participants | LB6 | Listing of All Urinalysis Data for Participants with Toxicities of Grade 2 or Higher | | SAC [1] |
| Electrod | ardiograms | | | | |
| 26 | All<br>Participants | EG6 | Listing of Abnormal ECG Findings | | SAC [1] |
| 27 | All<br>Participants | EG6 | Listing of All ECG Findings for Participants with an Abnormal Finding | | SAC [1] |
| 28 | All<br>Participants | EG4 | Listing of ECG Values of Potential Clinical Importance | | SAC [1] |
| 29 | All<br>Participants | EG4 | Listing of All ECG Values for Participants with any Value of Potential Clinical Importance | | SAC[1] |

| ICH : Lis | ICH : Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Vital Sig | jns | | | | |
| 30 | All<br>Participants | VS5 | Listing of Vital Signs of Potential Clinical Importance | | SAC [1] |
| 31 | All<br>Participants | VS5 | Listing of All Vital Signs for Participants with any Value of Potential Clinical Importance | | SAC [1] |
| Liver E | vent . | | | | |
| 32 | All<br>Participants | LIVER5 | Listing of Liver Monitoring/Stopping Event Reporting | | SAC[1] |
| 33 | All<br>Participants | МН3 | Listing of Medical Conditions for Participants with Liver Stopping Events | | SAC[1] |
| 34 | All<br>Participants | SAFE_L5 | Listing of Alcohol Intake at Onset of Liver Event | | SAC[1] |
| 35 | All<br>Participants | PKCL1X | Listing of Plasma Concentration Data for Participants with Liver Stopping Events | | SAC[1] |
| 36 | All<br>Participants | LIVER7 | Listing of Liver Biopsy Details | | SAC[1] |
| 37 | All<br>Participants | LIVER8 | Listing of Liver Imaging Details | | SAC[1] |

# 10.10.9. Other (non-ICH) Listings

| Julei (I | non-ICH) : Listing | 1 | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Pharma | cokinetic | | | | |
| 38 | PK | PKCL1X | Listing of DTG Plasma Pharmacokinetic Concentration-Time Data by Treatment | Please list all the concentration data including unscheduled. Repeat for all treatments and Parts. | SAC [1] |
| 39 | PK | PKCL1X | Listing of ABC Plasma Pharmacokinetic Concentration-Time Data by Treatment | Please list all the concentration data including unscheduled. Repeat for all treatments of Part 1. | SAC [1] |
| 40 | PK | PKCL1X | Listing of 3TC Plasma Pharmacokinetic Concentration-Time Data by Treatment | Please list all the concentration data including unscheduled. Repeat for all treatments and Parts. | SAC [1] |
| 41 | PK | PKPL1X | Listing of Derived DTG Plasma Pharmacokinetic Parameters by Treatment | Repeat for all treatments and Parts. | SAC [1] |
| 42 | PK | PKPL1X | Listing of Derived ABC Plasma Pharmacokinetic Parameters by Treatment | Repeat for all treatments of Part 1. | SAC [1] |
| 43 | PK | PKPL1X | Listing of Derived 3TC Plasma Pharmacokinetic Parameters by Treatment | Repeat for all treatments and Parts. | SAC [1] |
| Explora | itory | | | | |
| 44 | All<br>Participants | EXP_L1 | Listing of Palatability Questionnaire Results (Part 1, Treatment B Only) | | SAC[1] |
| 45 | All<br>Participants | EXP_L1 | Listing of Palatability Questionnaire Results (Part 2, Treatment E Only) | | SAC[1] |

# 10.11. Appendix 11: Example Mock Shells for Data Displays

Available upon request